CLINICAL TRIAL: NCT05887609
Title: A Phase II Evaluation of Maintenance Therapy Combination Mirvetuximab Soravtansine-gynx and Olaparib in Recurrent Platinum Sensitive Ovarian, Peritoneal, and Fallopian Tube Cancer
Brief Title: An Evaluation of Maintenance Therapy Combination Mirvetuximab Soravtansine and Olaparib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-0384.cc
Record Dates: First submitted 2023-05-10; First posted 2023-06-05 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Ovary Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — mirvetuximab soravtansine; olaparib

STUDY DESIGN:
Intervention Model Description: Single-arm, study design evaluating the maintenance therapy combination Mirvetuximab soravtansine-gynx and Olaparib in recurrent platinum-sensitive ovarian, peritoneal, and fallopian tube cancers. A six-patient safety lead in will occur, in which relevant the pharmaceutical company will be informed and included in safety evaluation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Lead In (Experimental)
  Interventions: Drug: Mirvetuximab Soravtansine-gynx; Drug: Olaparib
- Treatment (Experimental): All patients will receive MIRV at 5mg/kg AIBW administered through IV infusion on Day 1 of every 3-week cycle (Q3W).
  All patients will receive Olaparib at 300mg taken orally twice daily with or without food. Dosage and administration will follow current single-agent Olaparib package insert dosage and administration guidelines.
  Patients will continue to receive MIRV and Olaparib until PD, unacceptable toxicity, withdrawal of consent, or death, whichever comes first. If toxicity deems the patient to discontinue one drug, the patient may continue the other drug until PD, unacceptable toxicity, withdrawal of consent, or death, whichever comes first.
  Interventions: Drug: Mirvetuximab Soravtansine-gynx; Drug: Olaparib

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine-gynx — is an antibody-drug conjugate (ADC) that consists of a high affinity humanized monoclonal antibody against folate receptor α (FRα, the protein product of the folate receptor 1 [FOLR1] gene) that is conjugated to a cytotoxic maytansinoid by the hindered disulfide succinimidyl 4-(pyridine-2-yl)disulfanyl)-2-sulfo-butyrate linker (sulfo-SPDB).
  Other Names: IMGN853; MIRV
Drug: Olaparib — Olaparib is an inhibitor of poly (ADP-ribose) polymerase (PARP) enzymes, including PARP1, PARP2, and PARP3. PARP enzymes are involved in normal cellular functions, such as DNA transcription and DNA repair.

SUMMARY:
The Principal Investigator hypothesizes the combination of MIRV and Olaparib is an effective, and tolerable, maintenance therapy strategy in platinum sensitive recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision to sign and date the consent form
* Stated willingness to comply with all study procedures and be available for the duration of the study
* Be a woman aged ≥18 years of age
* Patients must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Patients must have a confirmed diagnosis of high-grade serous or endometrioid EOC, primary peritoneal cancer, or fallopian tube cancer
* Patients must have platinum-sensitive disease defined as radiographic progression greater than 6 months from last dose of prior platinum therapy (not inclusive of current/most recent platinum therapy)
* Patients must have had documented complete or partial response, or stable disease, as defined by RECIST 1.1, from last line of platinum therapy
* Patients must have available archival tissue block or slides to confirm FRalpha positivity
* Patients' tumor must have FRalpha high or medium expression
* Prior anticancer therapy:

  * Patients must have received at least one prior platinum-based chemotherapy regimen for platinum sensitive recurrent disease.
  * Most recent prior chemotherapy regimen must have consisted of at least 4 completed cycles and no more than 8 completed cycles
  * Most recent prior chemotherapy regimen must have been platinum based
  * Patients must have had testing for BRCA mutation (tumor or germline) and, if positive, must have received a prior PARP inhibitor as either treatment or maintenance therapy
  * Neoadjuvant +/- adjuvant therapies are considered 1 line of therapy
  * Maintenance therapy (eg, Bevacizumab, PARP inhibitors) will be considered part of preceding line of therapy (ie, not counted independently)
  * Therapy changed due to toxicity in the absence of progression will be considered part of the same line (ie, not counted independently)
  * Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance
  * Prior Bevacizumab use is allowed, but concurrent use with study combination is prohibited.
  * Cycle 1 Day 1 of trial therapy must be within 8 weeks of last dose of previous chemotherapy.
* Patients must have adequate hematologic, liver, and kidney function as defined as:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/µL)
  * Platelet count ≥ 100 x 109/L (100,000 µL)
  * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test
  * Aspartate aminotransferase (AST)(Serum Glutamic Oxaloacetic Transaminase (SGOT)) and alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x ULN unless liver metastases are present in which case they must be ≤ 5x ULN
  * Serum bilirubin ≤ 1.5 x ULN (patients with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 x ULN)
  * Serum albumin ≥ 2 g/dL

Exclusion Criteria:

* Patients with clear cell, mucinous, sarcomatous, low grade/borderline, germ cell, or sex-cord stromal type ovarian tumor
* Patients who have progressed through most recent chemotherapy regimen. Stable disease (SD) is permissible.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Patients with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions require ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and/or monocular vision
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to:

  * Uncontrolled major seizure disorder
  * Unstable spinal cord compression
  * Any psychiatric disorder that prohibits obtaining informed consent.
  * Active hepatitis B or C infection (whether or not on active antiviral therapy)
  * Immunocompromised patients, e.g., patient who are known to be serologically positive for human immunodeficient virus(HIV)
  * Active cytomegalovirus infection
  * Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to the first dose of MIRV
* Patients with a history of multiple sclerosis (MS) or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
* Patients with clinically significant cardiac disease including, but not limited to, any of the following

  * Myocardial infarction ≤ 6 months prior to first dose
  * Uncontrolled ventricular arrhythmia, recent (within 3 months)
  * Superior vena cava syndrome
  * Unstable angina pectoris
  * Uncontrolled congestive heart failure (New York Heart Association > class II)
  * Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
  * Uncontrolled cardiac arrhythmias
* Patients with a history of hemorrhagic or ischemic stroke within 6 months prior to enrollment
* Patients with a history of cirrhotic liver disease (Child-Pugh Class B or C)
* Patients with a previous clinical diagnosis of noninfectious interstitial lung disease (ILD) or Extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan , including noninfectious pneumonitis
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia
* Patients requiring use of folate-containing supplements (eg, folate deficiency)
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients with prior hypersensitivity to monoclonal antibodies (mAb)
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Women who are pregnant or breastfeeding, and who do not agree to use a highly effective contraceptive method(s) while on study drug and for at least 3 months after the last dose of MIRV and at least 6 months after the last dose of Olaparib. Females of childbearing potential must have a negative serum pregnancy test within 72 hours of study entry.
* Patients who received prior treatment with MIRV or other FRα- targeting agents
* Patients with duodenal stent or other GI disorder/defect that would interfere with absorption of oral medication

  * Includes patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Patients with known untreated or symptomatic central nervous system (CNS) metastases
* Patients with a history of other malignancy within 3 years prior to enrollment

  * Note: patients with tumors with a negligible risk for metastasis or death (eg, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible
* Prior known hypersensitivity reaction to study drugs and/or any of their excipients
* Minor or major surgical procedure within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Inability to comply with study and follow-up procedures
* Patients deemed otherwise clinically unfit for clinical trial per investigators discretion

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Be a woman aged ≥18 years of age
Enrollment: 53 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
To measure progression free survival (PFS) with the use of MIRV combined with Olaparib in women with recurrent platinum sensitive ovarian, peritoneal, and fallopian tube cancer. | Through study completion, average of 12 months
  PFS will be defined as the time from first dose of MIRV and Olaparib until investigator-assessed radiologic PD or death, whichever occurs first

SECONDARY OUTCOMES:
To evaluate safety and tolerability of MIRV combined with Olaparib by Adverse Events as measured by CTCAE v 5.0 | Through study completion, average of 12 months
  The team will use treatment-emergent adverse events (TEAEs) and laboratory test results, physical examination, or vital signs to determine AEs as described by CTCAE v5.0
Determine Overall Response Rate | Through study completion, average of 12 months
  Defined by confirmed best response of CR or PR as assessed by the investigator
Determine Duration of Response | Through study completion, average of 12 months
  Defined as the time from initial investigator-assessed response (CR or PR) until progressive disease (PD) as assessed by the investigator
Determine Overall Survival | Up to 5 years
  Defined as the time from first dose of MIRV and Olaparib until death

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Corr, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - University of Colorado Hospital, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Pennsylvania Health System, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - UPMC Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - University of Wisconsin - Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No